CLINICAL TRIAL: NCT04445766
Title: Efficacy and Complications of Microvascular Decompression - a Prospective Systematic Study of 115 Trigeminal Neuralgia Patients
Brief Title: Efficacy and Complications of Microvascular Decompression
Status: Completed | Type: Observational
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Lars Bendtsen, MD, PhD, Dr Med Sci, Danish Headache Center
Other Study IDs: H-16019808
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Trigeminal Neuralgia
Keywords: neurosurgery
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is a non-interventional prospective observational study in patients with trigeminal neuralgia that undergoes micovascular decompression. The aim is to evaluate the efficacy and complications 2 years after microvascular decompression

DETAILED DESCRIPTION:
The aim of this study is to prospectively evaluate effect and complications 2 years after MVD using independent assessors of outcome and complications.

Data of outcome and complications is collected prospectively based on based on standardized follow-up schemes and questionnaires. Patients were assessed by independent assessors before surgery and 3, 6, 12 and 24 months after surgery. Current pain level was evaluated according to VAS and BNI pain scale. Complications were evaluated by the assessors by a questionnaire and physical examination. All patients undergo a pre-surgical protocolized 3.0 Tesla MRI of the brain and brainstem.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Most give Signed informed Consent.
* Must fullfil the ICHD-3 beta diagnostic criteria for classical TN.Patients with purely paroxysmal TN and patients with TN with concomitant persistent facial pain will be included.
* If the ICHD-3 beta diagnostic criteria is fulfilled and if complete clinical history, neurological and physical examination and a 3.0 Tesla MRI do not raise any suspicion of another causative disease such as painful posttraumatic trigeminal neuropathy or symptomatic TN, subjects with sensory abnormalities detected at clinical neurological examination are also included.
* Has had a 3.0 Tesla MRI according to the trigeminal neuralgia protocol, prior to the surgical intervention.
* Semi-structured interview and neurological examination by the independent assessors prior to neurosurgical intervention.
* Has tried at least one, preferably two, sodium channel blocker (either carbamazepine or oxcarbazepine) before referral to neurosurgery.

Exclusion Criteria:

Subjects will be excluded if one of the following exclusion criteria is met:

* Psychiatric or mental illness or condition that might interfere with the ability of the patients to fill in the Informed Consent and questionnaires.
* Previous microvascular decompression as a treatment for trigeminal neuralgia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We consecutively evaluated patients with the diagnosis of TN seen at the Danish Headache Center (DHC), a tertiary medical referral centre for headache and facial pain. Patients who were treated with MVD at the Department of Neurosurgery were included in the study.
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Degree of pain relief 2 years after MVD | 2 years
  Barrow Neurological Institute pain intensity score (BNI)
Degree of complication rate 2 years after MVD | 2 years
  The frequency of predefined major and minor complications

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andersen ASS, Heinskou TB, Rochat P, Springborg JB, Noory N, Smilkov EA, Bendtsen L, Maarbjerg S. Microvascular decompression in trigeminal neuralgia - a prospective study of 115 patients. J Headache Pain. 2022 Nov 19;23(1):145. doi: 10.1186/s10194-022-01520-x. PMID 36402970